CLINICAL TRIAL: NCT05060198
Title: Open Label Randomized Study Evaluating the in Vivo Efficacies of Artemether-lumefantrine and Dihydroartemisinin-piperaquine in the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Children Under Five Years of Age in Western Kenya
Brief Title: Therapeutic Efficacy Study of AL and DP in Western Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenya Medical Research Institute (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Simon Kariuki, Malaria Branch Chief, Kenya Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2857
Record Dates: First submitted 2021-01-13; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Malaria,Falciparum
Keywords: Malaria; Kenya; Therapeutiic Efficacy; Artemether-lumefantrine; Dihydroartemisinin-piperaquine
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Artemether-lumefantrine (AL) (Active Comparator): Participants will be randomized to receive a standard weight-based regimen of artemether-lumefantrine (Coartem®, Novartis Pharmaceuticals Corporation, Missouri, USA). Children in the AL arm received two daily doses (morning and evening) orally, over 3 days (6 doses total at 0, 8, 24, 36, 48, and 60 hours post initial dose, administered with food or milk at the clinic and at home). To promote and evaluate adherence, study staff called parents in the evening to remind them to give the AL dose to the child and to bring the blister pack to the clinic the next day for confirmation.
  Interventions: Drug: Artemether-lumefantrine (AL)
- Dihydroartemisinin-piperaquine (DP) (Active Comparator): Participants will be randomized to receive a standard weight-based regimen of dihydroartemisinin-piperaquine (DuoCotexin®; Holley-Cotec Pharmaceuticals, Beijing, China). DP was administered once a day for three days (at 0, 24, and 48 hours, orally).
  Interventions: Drug: Dihydroartemisinin-piperaquine (DP)

INTERVENTIONS:
Drug: Artemether-lumefantrine (AL) — AL is the current first-line antimalarial in Kenya, per Kenya Ministry of Health.
  Other Names: Coartem
  Arms: Artemether-lumefantrine (AL)
Drug: Dihydroartemisinin-piperaquine (DP) — DP is the current second-line antimalarial in Kenya, per Kenya Ministry of Health.
  Other Names: Duocotexin
  Arms: Dihydroartemisinin-piperaquine (DP)

SUMMARY:
Artemether-lumefantrine (AL) was adopted as first-line antimalarial therapy in Kenya in 2006, and dihydroartemisinin-piperaquine (DP) as the second-line therapy in 2010. In order to monitor the efficacy and potential development of resistance of Plasmodium falciparum parasites to these two drugs, we will conduct an in-vivo study to monitor the efficacy of these antimalarial therapies.

A standardized World Health Organization (WHO) in-vivo efficacy study will be conducted in western Kenya among children 6-59 months of age with symptomatic, uncomplicated malaria visiting the out-patient department of hospitals and/or clinics in western Kenya.

In this study, 350 children will be randomly assigned to be treated with either AL or DP. Clinical, parasitologic, and hematologic parameters will be monitored over a 42-day follow-up period. Molecular analysis will be conducted to determine the frequency of markers of antimalarial resistance, and to differentiate recrudescence from reinfection. Results from this antimalarial drug efficacy study will be used to assist the Kenya national malaria control program (NMCP) in evaluating the national malaria treatment policy.

DETAILED DESCRIPTION:
Aim & Objectives

Aim: To assess the therapeutic efficacy of AL and DP for symptomatic, uncomplicated P. falciparum infections among children based on parasitologic, clinical, and hematologic parameters.

Objectives

i. To measure the clinical and parasitological efficacy of AL and DP among patients aged 6-59 months with symptomatic, uncomplicated P. falciparum malaria,

1. Primary efficacy endpoint: PCR-corrected parasitemia by day 42, the adequate clinical and parsitological response (ACPR)
2. Secondary efficacy endpoints:

   * Determine the proportion of children with early treatment failure (ETF) and late treatment failure (LTF) by determining the presence of parasitemia on days 3, 7, 14, 28, 35, and 42
   * To determine the frequency of existing molecular markers for drug resistance and identify new molecular markers
   * Evaluate drug concentration levels at day 7
   * Evaluate duration of malaria HRP2/pLDH RDT positivity after appropriate treatment with AL and DP

Design and Methodology Design: Randomized open-label clinical trial.

1. Study site. The study will be conducted at hospitals and/or clinics in western Kenya. This region of Kenya has some of the highest prevalence of malaria in Kenya. The decision of the site/s for each study will be determined prior to the initiation of each study and by criteria including: 1) sufficient number of children <5 years of age presenting to the site with symptomatic, uncomplicated malaria in the prior year, 2) ≥20 children presenting to the study site with symptomatic laboratory confirmed malaria per week, and 3) willingness of the staff to participate in the trial including the clinical and laboratory aspects.
2. Study population. The population of interest consists of patients aged 6-59 months diagnosed with symptomatic, uncomplicated P. falciparum malaria consulting at the study site, and whose parents or guardians give permission for study inclusion.
3. Intervention. Participants will be randomized to receive a standard weight-based regimen of: (1) artemether-lumefantrine (Coartem®, Novartis Pharmaceuticals Corporation, Missouri, USA) or (2) dihydroartemisinin-piperaquine (Duo-Cotecxin®, Holley-Cotec Pharmaceuticals, Beijing, China).
4. Consenting and Screening. Parents/guardians of patients presenting to the outpatient clinics with a clinical diagnosis of uncomplicated malaria will be approached by a team member and asked if they would be interested in joining the research study. The team member will explain the purpose and the procedures of the study, will review the inclusion and exclusion criteria with the parent/caregiver, and if the patient is eligible, and the patient/caregiver agrees, will then administer the consent to the parent/guardian.

   Study enrolment procedures:

   - The patient will be assigned a unique study identification number; this will be used to identify all forms and blood samples from that patient
   * Children will be evaluated by clinical staff for signs of febrile illness other than malaria, and signs of severe disease/ danger signs
   * Demographic and clinical data will be entered into a standardized form, including age, gender, axillary temperature, height, and body weight
   * A fingerprick will be performed to prepare a thick and a thin blood smear for microscopy, malaria RDT, hemoglobin determination by HemoCue®, and a filter paper blood for later PCR testing; the total blood volume collected will be <500 microliters.
   * Blood smear: The first thick smear will be stained with 10% Giemsa and quickly assessed for the presence of malaria parasitemia and an estimate of the parasite density.
5. Randomization & Blinding. Children will be block randomized to one of the study arms. The allocation will be blinded only to the microscopists reading the blood films.

Clinical Procedures.

1. After confirmation of enrolment:

   1. In order to easily identify patients in the community, digital photograph of both the child and parent/ guardian will be taken to verify the child's identity on repeat visits
   2. After randomization (day 0), each child will receive the (first) daily dose of study medication under direct observation and will be monitored for vomiting for 30 minutes. If a child vomits within 30 minutes of receiving their initial dose, the child will be retreated with the same dose of medication and observed for an additional 30 minutes. If vomiting continues, the child will be withdrawn from the study, and given rescue medication.
   3. If the child is taking AL, the parent will be given the evening dose to administer at home. Study personnel will attempt to confirm adherence by:

<!-- -->

1. Calling the parent/guardian twice to remind to dose the child
2. Request the parent/guardian to return with the blister pack so that a study member can visualize the number of doses remaining
3. Give the parent/guardian a reserve dose in the event that the child vomits the dose; request that the parent/guardian return the extra dose on day 7 to prevent administration of the extra dose.

b. Follow-up

1. Each child will return on days 1 and 2 for subsequent doses. Clinical reassessments will be made on days 1-3, 7, and then weekly until day 42 inclusive.
2. Patients will be advised to return on any day or night during the follow-up period if symptoms return and not to wait for scheduled visit days. We will call the parent/guardian of the child the day prior to a visit to remind them to come to the clinic. Patients who do not present to the study site for follow-up visits will be followed at home within 24 hours.
3. Parents will be reimbursed for transport per KEMRI/CDC guidelines for each visit to cover their travel expenses, and a long-lasting insecticide-treated bed net will be offered to the parent of each enrolled child at the time of enrollment.

   c. Blood samples.

   Blood films for parasite count will be obtained and examined on days 0, 2, 3, 7, 14, 21, 28, 35, and 42, on day 1 in case of sign/symptoms of severe malaria, and on any other day if the patient spontaneously returns with fever or worsening symptoms. Hemoglobin status will be measured on days 0, 7, 14, 28 and 42. A filter paper blood spot or blood collected in a microtainer tube (<1 ml blood) will be collected on day 7 to assess drug levels, and additionally on days 0, and after day 7 to assess parasite genotypes in the setting of late clinical failures; additional filter paper samples will be collected after day 3 in case of treatment failure and used to test for parasite species and polymorphism to distinguish between reinfection and recrudescence and for molecular markers of drug resistance as described below.

   Rescue Treatment.

   Patients with recrudescent infection or reinfection during the follow-up period will be treated with quinine. Patients with severe malaria will be referred to the hospital for in-patient treatment according to Kenya national guidelines (currently parenteral quinine or artesunate).

   Concomitant Treatment.

   Using standard clinic procedures, clinic personnel will administer supportive treatment to patients as necessary:

   • Antipyretics will be given for temperatures > 37.5C as per national policy.

   • Ferrous sulfate/ folate will be given to all children with hemoglobin <10 mg/dl as per national Integrated Management of Childhood Illness (IMCI) Guidelines

   • Anti-helminthics will be given to all children as per national IMCI Guidelines

   Study Endpoints

   Valid study end-points include treatment failure, completion of the follow-up period without treatment failure, loss to follow-up, withdrawal from study (voluntary or involuntary, and protocol violation). Loss to follow-up occurs when, despite all reasonable effort, an enrolled patient who does not attend the scheduled visits cannot be found within 3 days of their scheduled visit.

   Handling of Unexpected or Adverse Events.

   a. Identifying, managing and reporting adverse events. Existing data suggest that the drug combinations proposed in this study are safe. The combination of artemether-lumefantrine has been shown to be safe and highly efficacious. The combination of DHA-piperaquine has been shown to be safe, with mild adverse events, primarily gastrointestinal, headache, and mild QTc prolongation. Most severe allergic reactions would be expected to manifest within an hour of taking the dose. We will counsel parents to return immediately if their child develops a raised rash (i.e., urticaria) or difficulty breathing suggestive of a severe allergic reaction.

   b. Emergency Care. Mild adverse reactions will be noted in the case report form; no further action will be taken by study staff, except in the case of vomiting. For vomiting, the study medication will be re-administered according to the protocol. In the event of significant vomiting, initially ORS (oral rehydration solution) will be administered. If ORS is not tolerated, the patient will be referred to the hospital for management. In the case of any severe adverse reaction (e.g., difficulty breathing, convulsions, change in mental status), subjects will also be referred to hospital for management. Patients with signs of severe malaria, persistent vomiting or severe side effects will be referred to the hospital to receive parenteral therapy with quinine and relevant supportive treatments.

   c. Reporting adverse events. Any adverse event which is severe, unexpected, and possibly related to the research, as well as any unanticipated problems involving risks to subjects or others and any occurrences of serious or continuing non-compliance will be reported to the KEMRI and CDC IRB, according to their respective policies on incident reporting. Fatal outcomes will be reported within 2 days. A home visit will be conducted following the death of a child to assess the duration of illness, signs and symptoms of illness.

   Laboratory procedures: Polymerase Chain Reaction (PCR)

   In order to differentiate a recrudescence (same parasite strain) from reinfection (different parasite strain), a genotypic analysis based on merozoite surface protein-1 (msp1), merozoite surface protein 2 (msp2) and glutamate-rich protein (glurp) will be performed by PCR. Nested mutation-specific PCR, pyrosequencing or sequencing will be performed to analyze drug resistant mutations. We will investigate artemisinin resistance by evaluating mutations in the P. falciparum K-13 propeller gene, and potentially other genes including Pfcrt ,Pfmdr1.10 We plan to assess for the presence of these mutations in the western Kenyan parasite populations and characterize any potential new molecular markers as new information appears in the literature.

   Data analysis

   Data will be analyzed using two methods: survival analysis where children are included in the analysis until the last day before drop-out and a per-protocol analysis excluding all reinfections.

   The final analysis will include:

   - A description of the patients screened, and the distribution of the reasons for study exclusion.
   * A description of the patients included in the study.
   * The PCR corrected and uncorrected proportion of ETF, LCF, LPF, and ACPR in each treatment arm at day 28 and day 42 with 95% confidence intervals using survival analysis.
   * Frequency of side effects, severe malaria, anemia, and hospitalizations by treatment arm
   * The frequency of molecular markers for drug resistance

   Ethical Considerations

   The research will be conducted in compliance with the protocol, good clinical practice (GCP) guidelines, and all applicable regulatory requirements. Approvals will be obtained from KEMRI ERC and CDC IRB.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-59 months
2. Weight ≥ 5.0 kg
3. Axillary temperature ≥ 37.5C or history of fever in the past 24 hours
4. Hemoglobin ≥7 grams/deciliter at enrolment
5. Slide-confirmed mono-infection with Plasmodium falciparum and asexual parasite density between 2,000-200,000 parasites/μl
6. Live within the catchment boundaries of the study site (10km radius)
7. Able to swallow oral medication
8. Able and willing to comply with the protocol for the duration of the study
9. Able and willing to comply with the study visit schedule on days 2, 3, 7, 14, 21, 28, 35, and 42
10. Parent or caregiver has access to a phone and agrees to have study staff contact them for visit reminders during study period
11. Written informed consent provided by parent/guardian

Exclusion Criteria:

1. Presence of severe malaria or danger signs, including prostration, alteration in level of consciousness, respiratory distress, convulsions, or jaundice
2. Severe malnutrition according to WHO child growth standards (weight for age <3 standard deviations)
3. Known hypersensitivity to AL or DP
4. Use of antimalarials or other drugs with antimalarial activity in the last 2 weeks
5. General clinical condition necessitates hospitalization
6. Evidence of concomitant infections at the time of presentation
7. Plan to travel or leave the area within the next 3 months
8. Previously enrolled in this study

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 340 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Adequate clinical and parasitological response (ACPR) - AL | 28 days
  Absence of parasitemia on day 28 for AL, irrespective of axillary temperature, in patients who did not previously meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure.
Adequate clinical and parasitological response (ACPR) - DP | 42 days
  Absence of parasitemia on day 42 for DP, irrespective of axillary temperature, in patients who did not previously meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure.
Early treatment failure (ETF) | 3 days
  Danger signs or severe malaria on day 1, 2 or 3, in the presence of parasitemia;
  * Parasitemia on day 2 higher than on day 0, irrespective of axillary temperature;
  * Parasitemia on day 3 with axillary temperature ≥ 37.5 °C; and
  * Parasitemia on day 3 ≥ 25% of count on day 0.
Late clinical failure (LCF) - AL | 28 days
  Danger signs or severe malaria in the presence of parasitemia on any day between day 4 and day 28 for AL in participants who did not previously meet any of the criteria of early treatment failure; and
  • Presence of parasitemia on any day between day 4 and day 28 for AL with axillary temperature ≥ 37.5 °C in patients who did not previously meet any of the criteria of early treatment failure.
Late clinical failure (LCF) - DP | 42 days
  Danger signs or severe malaria in the presence of parasitemia on any day between day 4 and day 42 for DP in participants who did not previously meet any of the criteria of early treatment failure; and
  • Presence of parasitemia on any day between day 4 and day 42 for DP with axillary temperature ≥ 37.5 °C in patients who did not previously meet any of the criteria of early treatment failure.
Late parasitological failure (LPF) - AL | 28 days
  Presence of parasitemia on any day between day 7 and day 28 for AL with axillary temperature < 37.5 °C in patients who did not previously meet any of the criteria of early treatment failure or late clinical failure.
Late parasitological failure (LPF) - DP | 42 days
  Presence of parasitemia on any day between day 7 and day 42 for DP with axillary temperature < 37.5 °C in patients who did not previously meet any of the criteria of early treatment failure or late clinical failure.

SECONDARY OUTCOMES:
Change in hemoglobin over time | 42 days
  Change in hemoglobin
ACPR by baseline parasite density | 42 days
  Treatment efficacy stratified by baseline parasite density
Reinfection incidence rates and rate ratios by study arm, preventable fraction (AL) | 28 days
  Incidence rates calculated as number of reinfections per follow up period (28 days), by study arm; rate ratios by study arm, at 28 days; preventable fraction based on rate ratios, for 28 day follow up period.
Reinfection incidence rates and rate ratios by study arm, preventable fraction (DP) | 42 days
  Incidence rates calculated as number of reinfections per follow up period (42 days), by study arm; rate ratios by study arm, at 42 days; preventable fraction based on rate ratios, for 42 day follow up period.
Evaluate duration of malaria HRP2/pLDH RDT positivity after appropriate treatment with AL and DP | 42 days
  Using survival analysis, estimate median and end of follow up RDT positivity rate, by arm, baseline parasitemia, and in correlation with HRP2, LDH, and Aldolase lab values.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Kariuki, PhD, Principal Investigator — Kenya Medical Research Institute

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request
Supporting Information: Study Protocol, ICF
Time Frame: June 2021
Access Criteria: To be determined, depending on repository

REFERENCES:
- [Derived] Westercamp N, Owidhi M, Otieno K, Chebore W, Buff AM, Desai M, Kariuki S, Samuels AM. Efficacy of Artemether-Lumefantrine and Dihydroartemisinin-Piperaquine for the Treatment of Uncomplicated Plasmodium falciparum Malaria among Children in Western Kenya, 2016 to 2017. Antimicrob Agents Chemother. 2022 Sep 20;66(9):e0020722. doi: 10.1128/aac.00207-22. Epub 2022 Aug 29. PMID 36036611